CLINICAL TRIAL: NCT03680677
Title: Prospective Analysis of Frailty Phenotype Assessments to Optimize Treatment Strategies for Older Patients With Hematologic Malignancies
Brief Title: Frailty Phenotype Assessments to Optimize Treatment Strategies for Older Patients With Hematologic Malignancies
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 06718; 831340 (Other: U Penn IRB)
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Leukemia, Acute; MDS
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer Directed Therapy or Best Supportive Care: Cancer-directed therapy with intensive regimens, clinical trial, hypomethylating agent, hypomethylating agent combinations, targeted agents alone, or best supportive care
  Interventions: Other: Cancer-directed Therapy or Best Supportive Care; Diagnostic Test: Frailty Assessment
- Transplant: Bone marrow or peripheral blood graft (BMT) or CAR T-cell therapy
  Interventions: Procedure: Bone Marrow or Peripheral Blood Graft (BMT); Diagnostic Test: Frailty Assessment

INTERVENTIONS:
Procedure: Bone Marrow or Peripheral Blood Graft (BMT) — Patient receives bone marrow or peripheral blood graft (BMT) on or off protocol.
  Groups: Transplant
Other: Cancer-directed Therapy or Best Supportive Care — Cancer-directed therapy with intensive regimens ("7+3," Vyxeos, clofarabine, or similar), clinical trial, hypomethylating agent (azacitidine or decitabine), hypomethylating agent combinations (i.e. with venetoclax, sorafenib, enasidenib, ivosidenib, midostaurin, gilteritinib, or other targeted agent), targeted agents alone (i.e. enasidenib, ivosidenib, gilteritinib, midostaurin, etc.), or supportive care.
  Groups: Cancer Directed Therapy or Best Supportive Care
Diagnostic Test: Frailty Assessment — Frailty is the vulnerability of older adults to adverse health outcomes in response to illness and iatrogenic stressors.

SUMMARY:
The purpose of this research study is to determine if frailty assessments can be used to predict how well patients aged 60 years and older will do after chemotherapy, CAR T-cell therapy, or allogeneic stem cell transplant.

ELIGIBILITY:
Eligibility Criteria Arm A:

* Age 60 years or older.
* New diagnosis of Acute Leukemia or MDS, or suspected diagnosis.
* Able to consent to the study.

Eligibility Criteria Arm B:

* Age 60 years or older with a hematologic malignancy.
* Plan to undergo an allogeneic blood or marrow transplantation or CAR T-cell therapy.
* Able to consent to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts of patients will be included in this analysis.
  Arm A will include patients 60 years of age and older with a new diagnosis of either acute leukemia or MDS who are being evaluated either in the outpatient or inpatient hematologic malignancies department at the University of Pennsylvania.
  Arm B will include patients 60 years of age and older with a diagnosis of any hematologic malignancy being treated with cellular therapy including allogeneic blood or marrow transplantation or CAR T-cells.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Non-Relapse Mortality (NRM) in Frail, Pre-Frail, and Non-Frail patients | 1-month
  NRM will be defined as death without evidence of disease progression or relapse.

SECONDARY OUTCOMES:
NRM by Intensity of Treatment | 1-month and 6-month
  NRM of frail and pre-frail patients by intensity of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shannon McCurdy, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided